CLINICAL TRIAL: NCT04493775
Title: A Feasibility Study of Smartphone-based Brainwave Entrainment (BWE) Technology as a Novel Treatment for Chronic Pain
Brief Title: Smartphone-based Brainwave Entrainment (BWE) Technology in Chronic Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Helen Locke (Other)
Collaborators: University of Leeds (Other)
Responsible Party: Sponsor-Investigator, Helen Locke, Clinical Research Fellow, University of Manchester
Organization: University of Manchester (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NHS001675
Record Dates: First submitted 2020-07-21; First posted 2020-07-30 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-07

CONDITIONS: Chronic Pain
Keywords: Alpha rhythm; EEG phase synchronisation; Mobile applications; Pain perception; Pain management
MeSH Terms: conditions — Chronic Pain; Agnosia

STUDY DESIGN:
Masking Description: Neither the researcher delivering the intervention nor the participant will know the selected sequence at the start, however, it will not be possible for either the researcher or the participant to be completely blinded to the sequence once it is underway, given that the differences in duration of stimulation are likely to be quite apparent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Brainwave Entrainment — Alpha frequency visual and auditory stimulation delivered through a smartphone application, with the use of a virtual reality headset and earphones respectively.

SUMMARY:
Is brainwave entrainment a feasible tool for managing long-term pain in a patient population in the home-setting? Long-term pain affects 4 in 10 people in the UK and can impact on all aspects of life. Many people find that their pain is not well controlled on the treatments that are currently available, or they experience unpleasant side-effects from painkillers. There is therefore an urgent need for new safe and effective treatments for long-term pain.

One new approach to treatment is to target alpha brainwaves - rhythmic brain activity that is known to be associated with reduced pain. Alpha brainwaves can be increased by looking at flashing lights or listening to rhythmic sounds at the same rhythm as the brainwaves. This is known as "brainwave entrainment" (BWE) and can be delivered through a smartphone application.

The aim of this study is to test the suitability, acceptability and benefits of the brainwave entrainment smartphone application for people with long-term pain, and to inform the design of a future larger study.

The investigators aim to recruit 40 participants. Individuals may be eligible if they are over 18 years old and have suffered persistent pain for longer than 3 months. Participants will attend a 3-hour session in the laboratory in either Manchester or Leeds. They will undergo brainwave entrainment for different lengths of time whilst their brain activity and pain levels are recorded to determine the most effective "dose" of entrainment for that individual. They will then use the smartphone application at home 3 times a day for 4 weeks, and will complete pain, sleep, fatigue and quality of life questionnaires. At the end of the study, the investigators will conduct interviews to gain in-depth feedback. The total duration for each participant is around 7 weeks. This study is funded by a Leeds Cares Clinical Research Fellowship.

DETAILED DESCRIPTION:
Primary Question/Objective:

The principal research objectives are two-fold:

* Firstly, to understand the dose-response of alpha BWE.
* Secondly, to test the feasibility of using alpha BWE technology for managing chronic pain in the home environment and to inform the design of a future clinical trial.

Secondary Question/Objective:

* To identify any issues with recruitment or retention of participants.
* To test the acceptability and usability of the intervention.
* To test the acceptability of the outcome measures and methods of data collection.
* To gain an understanding of the effect size in order to calculate how many participants will be required for a future clinical trial.

STUDY DESIGN

Participants:

A total of 40 participants will be recruited from musculoskeletal, rheumatology and rehabilitation clinics in Leeds Teaching Hospitals National Health Service (NHS) Trust and Salford Royal NHS Foundation Trust.

Study Intervention and Procedures:

This is a two-stage feasibility study incorporating electroencephalography (EEG), quantitative outcome measures and qualitative interviews.

Project duration:

Each participant's involvement is estimated to last a minimum of 7 weeks (this may be longer depending on the availability of the participant to attend laboratory sessions).

Number of centres:

This study will be conducted across two sites: University of Manchester and University of Leeds. Two NHS sites will act as Participant Identification Centres (PICs): Leeds Teaching Hospitals Trust and Salford Royal NHS Foundation Trust.

Study design and procedures:

The project will be comprised of two studies: 1) a laboratory-based study followed by 2) a home-based study. All participants will be involved in both studies.

Potential participants may be approached and provided with a flyer and Participant Information Leaflet from musculoskeletal, rehabilitation and pain clinics at the two PICs, or may find out about the study from flyers placed in relevant NHS clinics or other relevant settings such as support groups. The participant will then contact the research team by phone or email on the contact details provided to discuss the study further, go through the screening process and arrange a convenient time for them to attend the laboratory if they wish to proceed.

Study 1:

Participants will attend either the University of Manchester laboratory in Salford Royal Hospital, or the University of Leeds laboratory in the School of Biological Sciences, University of Leeds, whichever is more convenient. They will be given opportunity to ask any questions before signing the consent forms. They will complete the following questionnaires:

* demographics form (5-10 mins)
* Pittsburg Sleep Quality Index (PSQI) (5-10 mins)
* Multidimensional Fatigue Index (MFI) (5-10 mins)
* EuroQol Five Dimensions (EQ-5D) (5-10 mins) Baseline EEG will be recorded for 7 minutes. The participant will then undergo 4 blocks of visual or auditory rhythmic stimulation (3 blocks of 10Hz visual stimulation lasting 5, 15 and 30 minutes and 1 block of non-entraining visual stimulation lasting 10 minutes) with 10-minute breaks in between as a wash-out period. EEG will continue to be recorded during these breaks. Participants will complete a Numerical Rating Scale (NRS) for pain intensity and unpleasantness before and after each block (<1 min). EEG will be recorded throughout stimulation.

Participants will then be introduced to the smartphone app, shown how to use it and given the opportunity to practice (30 mins). Participants will be provided with a smartphone with the BWE app pre-downloaded, a Virtual Reality (VR) headset and set of earphones to use for the duration of the study.

The estimated total laboratory time is 3 hours.

Study 2:

Participants will be asked to record NRS 3x a day and Brief Pain Index (BPI) short form (5-10 mins) 1x a day for 1 week at home to get baseline pain levels. After this period, they will be contacted by phone or email by a researcher to remind them to begin using the stimulation. They will then use the stimulation 3x a day for the specific duration that was identified as the optimum for them during the laboratory-based study (i.e. 5, 15 or 30 minutes, based on clinical pain ratings) for 4 weeks. They will record NRS for pain intensity and unpleasantness before and after each stimulation and BPI at the end of each day. This will be followed by a further week of baseline pain ratings with NRS 3x a day and BPI once a day.

Following this, the participant will attend the laboratory at a pre-arranged time to complete the following questionnaires:

* PSQI
* MFI
* EQ-5D (see study 1 for timings).

They will also participate in a semi-structured interview (<45 minutes) with a researcher. The interview will be based around a topic guide, however the semi-structured approach will allow for trajectories in the conversation according to any significant or relevant topics that may arise. The topic guide will be designed to:

1. Elicit participants' experiences of interacting with the app including factors affecting usability, adherence, the extent to which there has been any change in symptoms, any side effects and overall perceived usefulness and acceptability.
2. Explore any feasibility and process issues including factors affecting completion of outcome measures.

The interview will be audio-recorded and then transcribed verbatim with any identifiable data removed from the transcripts.

Recruitment:

Flyers advertising the study will be placed in relevant rheumatology, musculoskeletal and rehabilitation NHS clinics in Leeds and Manchester and in non-clinical settings (including support groups). Potential participants may be approached by clinicians in NHS clinics in the PICS, or they may contact the study team by telephone or email on the contact information provided on leaflets. Their eligibility for the study will be assessed by telephone. Participants will be provided with a verbal explanation and a Participant Information Leaflet (PIL) explaining the study, either in person or by email/post. They will have a minimum of 24 hours to decide whether to participate, at which point an initial meeting will be scheduled at a convenient date and time for the participant.

Written informed consent will be obtained from participants when they attend the laboratory for the initial meeting. Participants will have the opportunity to ask any further questions prior to consenting. A copy of the signed consent form will be given to the participant for their records and the original copy will be securely filed.

Randomisation:

All participants will receive the same intervention, however for study 1, the order in which the four sessions of stimulation (5, 15, 30 mins of alpha frequency and 10 mins of non-entraining stimulation) are delivered will be randomised using computer generated random numbers. A single research assistant who is not involved in delivery of the intervention will be responsible for the randomisation process. Neither the researcher delivering the intervention nor the participant will know the selected sequence at the start, however, it will not be possible for either the researcher or the participant to be completely blinded, given that the differences in duration of stimulation are likely to be quite apparent.

Statistical Analysis EEG data will be analysed using BrainVision Analyzer 2.0. Source localisation will be estimated using low resolution electromagnetic tomography (LORETA) using LORETA-KEY software. Appropriate statistical analysis will be carried out using SPSS software.

Interview findings will be explored with thematic content analysis using a Template Analysis approach. This involves the definition of a priori themes relevant to the research question. Two researchers will separately review and code an initial five transcripts based on the a priori themes, before coming together to organise the emerging themes into meaningful clusters and create an initial coding template by which to analyse the rest of the transcripts (modifying and revising the template as further themes emerge).

Sample Size:

The investigators aim to recruit a total of 40 participants who will take part in both work package 1 and 2. As a feasibility study, one of the key aims is to gain data on effect size in order to calculate sample size for a future clinical trial. Therefore, the sample size is based on previous studies as well as considering pragmatics such as funding, equipment and time available.

DATA MONITORING AND QUALITY ASSURANCE The study will be subject to the audit and monitoring regime of the Universities of Manchester and Leeds.

SAFETY CONSIDERATIONS AND ADVERSE EVENTS This study uses alpha frequency brainwave entrainment, which has no known significant side effects or risks. Therefore, the anticipated risk to participants is considered to be very low.

There are no anticipated risks to the researchers. There will be two-weekly debriefs with the whole research team to address any potential issues. There will be no lone-working for any team member.

ETHICAL and REGULATORY CONSIDERATIONS

Approvals:

The study will be conducted in full conformance with all relevant legal requirements and the principles of the Declaration of Helsinki, Good Clinical Practice (GCP) and the UK Policy Framework for Health and Social Care Research 2017. The study will be approved by NHS Research Ethics Committee and Health Research Authority prior to commencement.

Potential risks and burden to participants:

Due to the rhythmic flashing lights of the visual stimulation, individuals with a history of epilepsy or seizures will be excluded from the study, to mitigate the risk of triggering seizures. Those with sensitivity to flashing lights or a history of migraines or recurrent headaches will also be excluded. The brightness of the visual stimulation and the volume of auditory stimulation will be adjustable, to ensure it is comfortable. There are no known side effects from using this technology, however participants will be instructed to stop using it if they were to experience any adverse symptoms and to inform the research team.

Potential burden may arise from the inconvenience of attending the laboratory for face-to-face meetings. These have purposefully been kept to only 2 meetings to reduce this burden as much as possible. Data collection may be considered burdensome. Questionnaires at the beginning and end of the study will be completed with a researcher on hand to provide support. Although the NRS for pain takes seconds to complete, this will require participants to remember to record their pain scores three times a day. Participants will be provided with a clearly laid out booklet to assist them. Part of the feasibility aspect of this study is to assess how easy and acceptable the data collection measures are, so participants' feedback on the level of burden will be ascertained in the final interview and will guide future study design. Participants may perceive some burden from the final interview. It is not anticipated that the content will be upsetting for participants, however it is recognised that potentially sensitive topics may arise, including discussion of chronic pain and other symptoms. Participants will be informed that they do not have to answer any questions that they are uncomfortable with and they may leave the interview at any time without needing to give a reason.

ELIGIBILITY:
Inclusion Criteria:

* adults over the age of 18 years (there is no upper age limit as we would want the intervention to be as inclusive as possible)
* clinically significant non-cancer-related chronic pain (for which they have sought medical input) for more than three months' duration
* willing and able to consent to taking part.

Exclusion Criteria:

* any history or first-degree relative history of epilepsy or convulsions/seizures
* discomfort with flashing lights
* history of recurrent headaches or migraines
* participants who have difficulty understanding verbal or written English, or who have cognitive or mental health problems that would prevent them being able to provide written informed consent
* planned intervention (surgery, new medications or treatments) during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Numerical pain ratings (NRS) | 2 years
  0-10 where 0 = no pain and 10 = worst pain. To indicate whether there is a dose-related change in efficacy of BWE.
Qualitative data from semi-structured interviews | 2 years
  This will answer key feasibility questions to enable planning of a future clinical trial. This will include information on acceptability and usability of the intervention, feedback on the outcome measures used, engagement with the research, process issues including recruitment, and the extent to which they felt the intervention improved their pain.

SECONDARY OUTCOMES:
Electroencephalography data | 1 year
  Alpha frequency across all scalp electrodes (64 channel) recorded during rest and during alpha brainwave entrainment.
Pittsburgh sleep quality index (PSQI) | 2 years
  9 item questionnaire. The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Multidimensional Fatigue Inventory (MFI) | 2 years
  20 item questionnaire with each item scored from 1-5. Higher scores indicate a higher fatigue level.
EuroQol - 5 dimensions (EQ-5D) | 2 years
  Two components. 1. Health state description, five indicators whereby higher scores indicate better health in the last 24 hours. 2. Visual analogue scale 0-100 whereby 100 = best health imaginable and 0 = worst health imaginable.
Brief Pain Inventory (BPI) | 2 years
  Questionnaire with two categories: Pain Intensity (worst, least, on average, and currently) and Pain Interference (mood, work, general activity, walking, relationships, enjoyment of life, and sleep). Each category is rated 0-10. 10 = excruciating pain intensity and a complete interference in their life.

CONTACTS AND LOCATIONS:
Overall Officials: Jones, Principal Investigator — University of Manchester
Locations (2):
- United Kingdom (2):
  - University of Manchester, Manchester, Lancashire
  - University of Leeds, Leeds, West Yorkshire

IPD SHARING:
Plan to Share IPD: No